CLINICAL TRIAL: NCT03496038
Title: Trans-crestal Sinus Floor Elevation in Implant Therapy: A Randomized Controlled Clinical Trail With Parallel Group Design: L-PRF Compared With DBBM
Brief Title: Transcrestal Lateral Sinus Floor Elevation in Implant Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Dentsply International (Industry)
Responsible Party: Principal Investigator, Drs. Simone Cortellini, Clinical and Research Associate, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cortellini60096
Record Dates: First submitted 2018-03-19; First posted 2018-04-12 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Edentulous; Alveolar Process, Atrophy
MeSH Terms: conditions — Mouth, Edentulous; Atrophy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leukocyte and Platelet Rich Fibrin (L-PRF) (Experimental): For the test group the sub-sinus cavity will be filled with Leukocyte en Platelet Rich Fibrin (L-PRF).
  Before starting the surgery, 8 tubes (9 ml) of venous blood will be collected from the patients. A centrifugation standard L-PRF protocol will be followed followed (12 minutes centrifugation, 2700 rpm/408g RCF).
  After full centrifugation of the tubes, the L-PRF clots will be removed from the tubes using surgical tweezers. The clots will be thereafter gently compressed into membranes using a sterile metal box (Xpression, Intra-Lock, Florida, USA).
  Interventions: Procedure: L-PRF
- Deproteinized Bovine Bone Mineral (DBBM) (Active Comparator): For the test group the sub-sinus cavity will be filled with deproteinized bovine bone mineral (DBBM). The product used will be a xenograft (Bio-Oss Small particles, Geistlich AG, Wolhusen, Switzerland).
  Interventions: Procedure: DBBM

INTERVENTIONS:
Procedure: L-PRF — The use of the L-PRF as graft material for sinus augmentation procedure will be analysed
  Arms: Leukocyte and Platelet Rich Fibrin (L-PRF)
Procedure: DBBM — The use of bovine xenograft as graft material for sinus augmentation procedure will be analysed
  Arms: Deproteinized Bovine Bone Mineral (DBBM)

SUMMARY:
This is a non-inferiority study to evaluate whether L-PRF achieves similar or perhaps better results in bone gain, compared with "the golden standard" DBBM, after trans-crestal sinus floor elevation.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial with parallel group design. A total of 40 patients, needing transcrestal sinus lift (T), will be enrolled.

Under local anesthesia, the required T and implant placement will be performed and ISQ values will be recorded. Afterwards a CBCT will be taken for control. Randomization will be performed by computer generated random codes, using random permuted blocks with a block size of 4 to avoid uneven splits and minimization for the key prognostic factors RBH. Allocation will be concealed to the surgeons at completion of the common part of treatment, by opening an opaque envelope. At the same time an oral implant(s) will be inserted in the augmented area.

After 6 months a CBCT will be taken for control of the bone healing and the measurements of the newly formed bone. The abutment will be placed on top of the osseo-integrated implant(s) under local anesthesia. ISQ values will be recorded. Follow-up will be till 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Need for T and oral implant placement.
* RBH >3mm

Exclusion Criteria:

* Unlikely to be able to comply with the study procedures, as judged by the investigator
* Untreated periodontal disease
* Unfavorable plaque control
* Known or suspected current malignancy
* History of chemotherapy within 5y prior to study
* History of radiation on the head and neck region
* History of other metabolic bone diseases
* Need for systemic corticosteroids
* Current or previous use of intravenous/oral bisphosphonates
* Present alcohol and/or drug abuse
* Involvement in the planning and conduct of the study
* Psychiatric disorders which do not allow a normal treatment outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Volumetric bone regeneration en volumetric change | 6 and 12 months
  Amount of bone formation in healing period after trans-crestal sinus floor elevation and implant placement and after healing, measured on CBCT images.
  Following a healing period of 6 and 12 months a CBCT will be taken to measure the height and width of the newly formed bone and compare it to the initial CBCT. A 3-D volumetric analysis of the amount of gained bone is conducted with MeVisLab software.
Linear bone regeneration en lineair change | 6 and 12 months
  Amount of bone formation in healing period after trans-crestal sinus floor elevation and implant placement and after healing, measured on CBCT images.
  Following a healing period of 6 and 12 months a CBCT will be taken to measure the height and width of the newly formed bone and compare it to the initial CBCT. 2-D measurement will be performed.

SECONDARY OUTCOMES:
Implant stability based on resonance frequency | 6 months
  Measurements of the implant stability via Osstell ISQ implant stability device. At implant placement and abutment connection a measurement via Osstell ISQ implant stability device will be done.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No